CLINICAL TRIAL: NCT04000984
Title: Investigating the Beneficial Effects of Mindfulness-based Training on Neuropsychological Outcomes in Mild Cognitive Impairment
Brief Title: Beneficial Effects of Mindfulness-based Training on Neuropsychological Outcomes in Mild Cognitive Impairment
Acronym: MEDIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Singapore General Hospital (Other)
Collaborators: Duke-NUS Graduate Medical School (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: 2015/3149
Record Dates: First submitted 2019-05-06; First posted 2019-06-27 (Actual); Last update posted 2020-03-27 (Actual); Status verified 2020-03

CONDITIONS: Mild Cognitive Impairment
Keywords: Mindfulness; Cognitive Rehabilitation
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Cognitive Training

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to receive either the treatment intervention, Mindfulness-Based Intervention, compared against an active control, the Cognitive Rehabilitation Training in parallel and both groups will also be compared against a passive control group, the Treatment as Usual, where no intervention takes place.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Research Assistants who perform the pre- and post-assessments will not be privy to the group assignment of the participants and will not be involved in the data collection process during the duration of the intervention weeks.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Mindfulness-Based Intervention (Experimental): Participants in this arm will complete baseline and follow-up visits (approximately 3-months after) and Mid-intervention safety checks. They will attend the in the Mindfulness-Based Training program that will meet weekly for 8 weeks. Each session will last approximately one-and-a-half hours.
  Interventions: Behavioral: Mindfulness Based Training (MBT) Program
- Cognitive Rehabilitation Training (Active Comparator): Participants in this arm will complete baseline and follow-up visits (approximately 3-months after) and Mid-intervention safety checks. They will attend the Cognitive Rehabilitation program that will meet weekly for 8 weeks. Each session will last one-and-a-half hours.
  Interventions: Behavioral: Cognitive Rehabilitation Training
- Treatment As Usual (No Intervention): Participants in the Treatment As Usual group were only required to attend baseline and follow-up visits (approximately 3-months after) and Mid-intervention safety checks. Participants in this group will not receive an intervention for the duration of the study. They received treatment as usual which is 6 months to 1-year follow up visits with their attending neurologist of psychologist.

INTERVENTIONS:
Behavioral: Mindfulness Based Training (MBT) Program — Participants in the MBT program will meet weekly for 8 weeks. Each session will last one-and-a-half hours. Mindfulness, defined as caring moment-to-moment awareness, will be cultivated through the teaching and formal practice of sitting and walking meditation, body scan, and mindful movement (e.g. yoga). Participants will also be taught how to practice mindfulness informally when eating, engaging in pleasurable activities and through interactions with others. Participants will be encouraged to practice approximately 30 minutes a day, and will be provided handouts as well as guided audio recordings of formal practices taught in session to aid their practice at home.
  Other Names: MBT
  Arms: Mindfulness-Based Intervention
Behavioral: Cognitive Rehabilitation Training — Participants in the CRT program will meet weekly for 8 weeks. Each session will last one-and-a-half hours. The 8 week-program will consist of the following components: (i) identifying and working on at least one personal rehabilitation goal related to everyday life that is associated with cognitive difficulties; (ii) reviewing and building on the use of practical memory strategies, and or introducing and teaching the use of a new strategy or memory aid; (iii) introducing techniques for learning new information and associations, identifying the preferred strategy, and encouraging the application of this strategy in daily life; (iv) providing practice in maintaining attention and concentration; and (v) exploring current ways of coping with stress and anxiety as well as providing relaxation techniques to help aid with coping (Clare, 2007). Participants will be provided with instructional hand-outs as well as logs to record, monitor and evaluate their progress.
  Other Names: CRT
  Arms: Cognitive Rehabilitation Training

SUMMARY:
This study evaluates the effects of Mindfulness-based Interventions (MBI) on the neuropsychological profile of individuals with mild cognitive impairment (MCI). It will also investigate changes in fMRI activity, such as resting-state functional connectivity networks and changes in activity in attention networks in task-related fMRI using graph theory analysis after Mindfulness-based Interventions. Participants will be randomly assigned to receive either the Mindfulness-Based Intervention, Cognitive Rehabilitation Training or Treatment as Usual as the passive control group comparison.

DETAILED DESCRIPTION:
As the population of Singapore ages rapidly, cognitive decline associated with both normal aging and disease is becoming a frequently encountered health challenge. In our proposed study, we will investigate the effects of mindfulness-based interventions (MBI), which have shown significant promise in halting and even reversing age-related cognitive impairment. MBI enhances the quality and frequency of mindfulness, defined as a mental state achieved by focusing one's attention and awareness on the present moment, while calmly acknowledging and accepting one's feelings, thoughts, and bodily sensations. In this study, we will administer a standardized MBI program or Cognitive Rehabilitation Therapy to a group of 60 patients diagnosed with mild cognitive impairment (MCI), a condition marked by deficits in language, memory and attention that often leads to dementia; an additional 30 patients will be assigned to the control group. There will be 3 runs with 30 persons per run; each group will have 10 randomly assigned participants. By comparing the 3 groups across the 3 runs, we seek to test the following hypotheses: 1) MBI will result in significantly greater improvements in neuropsychological testing outcomes across multiple cognitive domains, including attention, memory, language and processing speed, 2) MBI will strengthen cortical connectivity as measured by functional magnetic resonance imaging (fMRI), and 3) MBI will lead to changes in fMRI activation on a test of facets of attention. Neuropsychological testing will take place in SGH, while fMRI and EEG scanning will take place in the Center for Cognitive Neuroscience at Duke-NUS. Both the MBI and CRT will be facilitated by trained personnel. Our proposed experiment comprises one of the most comprehensive interrogations of the effects of MBT on patients to date, and if successful, could rapidly translate into a program with both clinical and economic impact.

ELIGIBILITY:
Inclusion Criteria:

1. Fluent in English
2. Mild Cognitive Impairment: Fulfill Diagnostic and Statistical Manual of Mental Disorders version five (DSM-V) diagnostic criteria for Minor Neurocognitive Disorder
3. MMSE score = 20-30
4. Clinical Dementia Rating Score (CDR) = 0.5
5. Age: ≤75 years

Exclusion Criteria:

1. Presence of major neurological conditions such as epilepsy, stroke, Parkinson's Disease and or brain injury
2. Presence of major psychiatric conditions such as major depression or schizophrenia
3. Unsuitability for fMRI scanning (e.g. pacemakers, metallic implants, claustrophobia)
4. Unable to give or no consent available
5. Left-handed participants may take part in the study but will not undergo fMRI scanning

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2019-12-01 (Actual)

PRIMARY OUTCOMES:
Change in Attention | 10 minutes
  The RBANS Attention Index is a composite of the Digit Span and Coding subtests. This index is a measure of simple auditory registration and visual scanning and processing speed. Low scores on this index indicate difficulties with basic attention processes and speed of information processing.
Change in Immediate Memory | 10 minutes
  The RBANS Immediate Memory Index is composite of the learning (immediate) trials of the Story Memory and List Learning subtests. This index is a measure of initial encoding and learning complex and simple verbal information. Low scores on this index indicate difficulties with verbal learning.
Change in Delayed Memory | 30 minutes
  The RBANS Delayed Memory Index is a composite of the Story Memory Recall, List Learning Recall, List Learning Recognition, and Figure Recall subtests. This index is a measure of delayed recall and recognition for verbal and visual information. Low scores on this index indicate difficulties with recognition and retrieval of information from long-term memory stores.
Change in Processing Speed: Colour Trails 1 and 2 | 10 minutes
  Speed of cognitive processing and executive functioning is measured by the total time taken to complete each task.
Chang in Mindfulness Awareness and Attention Scores | An average of 3 months
  Dispositional Mindfulness and present-centered attention-awareness in everyday experience is measured with this scale. This instrument focused on the absence of attention to and awareness of present experience, and operationalized mindfulness as a single construct.

SECONDARY OUTCOMES:
Change in Subjective Quality of Life: Short-Form 36 | An average of 3 months
  Short-Form 36 (SF-36) is a 36-item self-report survey of health, including physical and mental health, with 8 scaled scores, each ranging from a minimum of 0 to max 100. Total score is the mean of all the subscales.
  Physical functioning : 10 items; Role functioning/physical : 4 items; Role emotional: 3 items; Energy/fatigue: 4 items; Mental Health: 5 items; Social functioning: 2 items; Body pain: 2 items; General health : 5 items; Reported health transition: 1 item.
Change in Subjective measures of Sleep quality: Insomnia Severity Index | Two weeks
  Insomnia Severity Index (ISI) evaluates an individual's level of tendency for insomnia on a 7-item questionnaire, scoring in total from 0 to 28. Scores above 15 indicates moderate severity of clinical insomnia while scores above 22 are indicative of severe clinical insomnia. ISI internal consistency was excellent for population samples both in the community and clinical samples as well, (Cronbach α of 0.90 and 0.91 respectively).
Change in Subjective measures of Sleep quality: Pittsburgh Sleep Quality Index Score | One month
  Pittsburgh Sleep Quality Index Score (PSQI) is a 19-item self-rated questionnaire for evaluating subjective sleep quality over the previous month. The PSQI has a sensitivity of 89.6% and specificity of 86.5% for identifying cases with sleep disorder, using a cut-off score of 5.
  The first 4 items are open questions, whereas items 5 to 19 are rated on a 4-point Likert scale. Individual items scores yield 7 components. A total score, ranging from 0 to 21, is obtained by adding the 7 component scores. A score of 5 and above suggests poor sleep quality. A decrease in PSQI score following intervention would reflect and improvement of sleep quality.
Imaging measures (structural): change in orbitofrontal cortex volume | 6 minutes
  The change in the volume of orbitofrontal cortex (OFC) is assessed through structural MRI brain scans - Participants will have their baseline fMRI scan before the start of their participation in the intervention and after the end of the intervention.
Change in functional imaging measures: Resting state | 10 minutes
  During two rsfMRI scans, subjects are imaged over several minutes while their eyes are open, but without performing any explicit task. The resting state scan will show only a fixation cross on the screen in order to minimize the cognitive processing involved while decreasing head movement and sleepiness in the scanner.
  Mindfulness predisposition is measured with the use of traditional connectivity analysis as well as a newer method: graph theory analysis for task ready state in Dynamic Functional Connectivity. These data are extracted by decomposing the time-varying signal during resting periods into independent, intrinsically connected networks.

CONTACTS AND LOCATIONS:
Overall Officials: Kinjal Doshi, PhD, Principal Investigator — Singapore General Hospital; Julian Lim, PhD, Principal Investigator — Duke-NUS Graduate Medical School
Locations (1):
- Singapore General Hospital, Singapore, Singapore

REFERENCES:
- [Background] Brier MR, Thomas JB, Fagan AM, Hassenstab J, Holtzman DM, Benzinger TL, Morris JC, Ances BM. Functional connectivity and graph theory in preclinical Alzheimer's disease. Neurobiol Aging. 2014 Apr;35(4):757-68. doi: 10.1016/j.neurobiolaging.2013.10.081. Epub 2013 Oct 18. PMID 24216223
- [Background] Bullmore E, Sporns O. Complex brain networks: graph theoretical analysis of structural and functional systems. Nat Rev Neurosci. 2009 Mar;10(3):186-98. doi: 10.1038/nrn2575. Epub 2009 Feb 4. PMID 19190637
- [Background] Dai Z, He Y. Disrupted structural and functional brain connectomes in mild cognitive impairment and Alzheimer's disease. Neurosci Bull. 2014 Apr;30(2):217-32. doi: 10.1007/s12264-013-1421-0. Epub 2014 Apr 15. PMID 24733652
- [Background] Dinges DF, Pack F, Williams K, Gillen KA, Powell JW, Ott GE, Aptowicz C, Pack AI. Cumulative sleepiness, mood disturbance, and psychomotor vigilance performance decrements during a week of sleep restricted to 4-5 hours per night. Sleep. 1997 Apr;20(4):267-77. PMID 9231952
- [Background] Fox MD, Raichle ME. Spontaneous fluctuations in brain activity observed with functional magnetic resonance imaging. Nat Rev Neurosci. 2007 Sep;8(9):700-11. doi: 10.1038/nrn2201. PMID 17704812
- [Background] Fox MD, Snyder AZ, Vincent JL, Raichle ME. Intrinsic fluctuations within cortical systems account for intertrial variability in human behavior. Neuron. 2007 Oct 4;56(1):171-84. doi: 10.1016/j.neuron.2007.08.023. PMID 17920023
- [Background] Gard T, Holzel BK, Lazar SW. The potential effects of meditation on age-related cognitive decline: a systematic review. Ann N Y Acad Sci. 2014 Jan;1307:89-103. doi: 10.1111/nyas.12348. PMID 24571182
- [Background] Gauthier S, Reisberg B, Zaudig M, Petersen RC, Ritchie K, Broich K, Belleville S, Brodaty H, Bennett D, Chertkow H, Cummings JL, de Leon M, Feldman H, Ganguli M, Hampel H, Scheltens P, Tierney MC, Whitehouse P, Winblad B; International Psychogeriatric Association Expert Conference on mild cognitive impairment. Mild cognitive impairment. Lancet. 2006 Apr 15;367(9518):1262-70. doi: 10.1016/S0140-6736(06)68542-5. PMID 16631882
- [Background] He X, Qin W, Liu Y, Zhang X, Duan Y, Song J, Li K, Jiang T, Yu C. Abnormal salience network in normal aging and in amnestic mild cognitive impairment and Alzheimer's disease. Hum Brain Mapp. 2014 Jul;35(7):3446-64. doi: 10.1002/hbm.22414. Epub 2013 Nov 12. PMID 24222384
- [Background] Huckans M, Hutson L, Twamley E, Jak A, Kaye J, Storzbach D. Efficacy of cognitive rehabilitation therapies for mild cognitive impairment (MCI) in older adults: working toward a theoretical model and evidence-based interventions. Neuropsychol Rev. 2013 Mar;23(1):63-80. doi: 10.1007/s11065-013-9230-9. Epub 2013 Mar 8. PMID 23471631
- [Background] Kilpatrick LA, Suyenobu BY, Smith SR, Bueller JA, Goodman T, Creswell JD, Tillisch K, Mayer EA, Naliboff BD. Impact of Mindfulness-Based Stress Reduction training on intrinsic brain connectivity. Neuroimage. 2011 May 1;56(1):290-8. doi: 10.1016/j.neuroimage.2011.02.034. Epub 2011 Feb 18. PMID 21334442
- [Background] Koepsell TD, Monsell SE. Reversion from mild cognitive impairment to normal or near-normal cognition: risk factors and prognosis. Neurology. 2012 Oct 9;79(15):1591-8. doi: 10.1212/WNL.0b013e31826e26b7. Epub 2012 Sep 26. PMID 23019264
- [Background] Lim J, Dinges DF. Sleep deprivation and vigilant attention. Ann N Y Acad Sci. 2008;1129:305-22. doi: 10.1196/annals.1417.002. PMID 18591490
- [Background] Manly JJ, Tang MX, Schupf N, Stern Y, Vonsattel JP, Mayeux R. Frequency and course of mild cognitive impairment in a multiethnic community. Ann Neurol. 2008 Apr;63(4):494-506. doi: 10.1002/ana.21326. PMID 18300306
- [Background] Mcbee, L. (2008) Mindfulness-based elder care. New York: Springer.
- [Background] Sun Y, Lim J, Kwok K, Bezerianos A. Functional cortical connectivity analysis of mental fatigue unmasks hemispheric asymmetry and changes in small-world networks. Brain Cogn. 2014 Mar;85:220-30. doi: 10.1016/j.bandc.2013.12.011. Epub 2014 Jan 21. PMID 24463002
- [Background] Tang YY, Ma Y, Fan Y, Feng H, Wang J, Feng S, Lu Q, Hu B, Lin Y, Li J, Zhang Y, Wang Y, Zhou L, Fan M. Central and autonomic nervous system interaction is altered by short-term meditation. Proc Natl Acad Sci U S A. 2009 Jun 2;106(22):8865-70. doi: 10.1073/pnas.0904031106. Epub 2009 May 18. PMID 19451642
- [Background] Tschanz JT, Welsh-Bohmer KA, Lyketsos CG, Corcoran C, Green RC, Hayden K, Norton MC, Zandi PP, Toone L, West NA, Breitner JC; Cache County Investigators. Conversion to dementia from mild cognitive disorder: the Cache County Study. Neurology. 2006 Jul 25;67(2):229-34. doi: 10.1212/01.wnl.0000224748.48011.84. PMID 16864813